CLINICAL TRIAL: NCT04060511
Title: A Phase 1, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of HS-10342 in Patients With Advanced Solid Tumor
Brief Title: A Study of HS-10342 in Patients With Advanced Solid Tumor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10342-101
Record Dates: First submitted 2019-08-15; First posted 2019-08-19 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
Keywords: CDK4/6 inhibitor, advanced solid tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS-10342 (Experimental): Each subject will receive a single dose(C0) of HS-10342 and then repeat doses(C1, C2…) for 28-day cycles. Participants may continue on study drug until disease progression, unacceptable toxicity, or other withdrawal criteria is met.
  Interventions: Drug: HS-10342

INTERVENTIONS:
Drug: HS-10342 — HS-10342 either 25mg, 50mg, 100mg, 150mg, 200mg given orally, QD or 50mg, 100mg, 150mg, 200mg, 250mg, 275mg given orally, BID

SUMMARY:
HS-10342 is a small molecular, oral potent, selective CDK4/6 inhibitor. The purpose of this study is to investigate the safety/tolerability and the pharmacokinetic profile of HS-10342 in Chinese advanced solid tumor patients. Preliminary efficacy will be also investigated in this study.

DETAILED DESCRIPTION:
This is a phase 1, multicenter study to evaluate the safety, tolerability, pharmacokinetics and efficacy of HS-10342 in patients with advanced solid tumor by using a "3+3" dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Pathologically confirmed solid tumor and failed from all standard treatment.
  2. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
  3. Eastern Cooperative Oncology Group (ECOG) performance status: 0-1.
  4. Life expectancy ≥ 3 months.
  5. Adequate function of major organs meets the following requirements:

     * Neutrophils ≥ 1.5×10^9/L
     * Platelets ≥ 90×10^9/L
     * Hemoglobin ≥ 90g/L
     * Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
     * ALT and AST ≤ 2.5 × ULN
     * Cr ≤ 1.5 × ULN
     * Left ventricular ejection fraction (LVEF) ≥ 40%
  6. Good compliance of patient by physician's judgement.
  7. . Signed and dated informed consent.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

  1. Previously received therapy of anti-tumor agent targeting at CDK4/6.
  2. Less than 3 weeks from the last cell-toxicity chemotherapy, less than 6 weeks from last mitomycin or nitrosamine therapy
  3. Less than 3 weeks from any other anti-tumor therapy (including targets therapy, immunotherapy or other approved therapy)
  4. Less than 4 weeks from large area radiotherapy.
  5. Less than 7 days from any CYP3A4 strong inhibitor, strong inducer or a narrow window of medicine or food for CYP3A4 sensitive substrate.
  6. Having joined in other clinical trials within 4 weeks.
  7. Brain metastasis (well-controlled/well-treated brain metastasis by physician's judgement is allowed).
  8. Existing abnormal CTCAE≥grade 2 resulted from previous treatment(except grade 2 alopecia).
  9. Uncontrollable pleural effusion or ascites.
  10. Inability to swallow, intestinal obstruction or other factors affecting the administration and absorption of the drug.
  11. History of serious allergy events or known being allergy constitution, or have a history of allergies to the drug components of this regimen.
  12. Patients with active infection.
  13. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation.
  14. History of uncontrollable cardiac dysfunction, include(1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction Less than 6 moths (4) other cardiac dysfunction (judged by the physician), such as any degree of heart block or QTc prolongation, QT interval corrected by Fridericia method(QTcF) >450 ms(men) or >470 ms(women); (5)any cardiac or nephric abnormal ≥ grade 2 found in screening.
  15. Males and females of reproductive potential who are unwilling to use an "effective", protocol specified method(s) of contraception during the study.
  16. Pregnant women, women who are breastfeeding or who believe they may wish to become pregnant during the course of the study.
  17. History of neuropathy or dysphrenia, including epilepsy and dementia
  18. Determined by the physician, any coexisting disease might lead to life threatening complications or avoid the patients from accomplishing the treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Eligibility is based on gender
Enrollment: 17 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicity and Maximum Tolerated Dose of HS-10342. | 5 weeks
  The maximum-tolerated dose (MTD) will be defined as the maximum dose level at which no more than one out of three subjects experience a dose-limiting toxicity (DLT) within the 5 week after the first dose.

CONTACTS AND LOCATIONS:
Overall Officials: Binhe Xu, MD, Principal Investigator — Cancer Hosptial, Chinese Academy of Medical Sciences; Herui Yao, MD, Principal Investigator — Second Affiliated Hospital, Sun Yat-Sen University; Qiang liu, MD, Principal Investigator — Second Affiliated Hospital, Sun Yat-Sen University; Yongmei Yin, MD, Principal Investigator — Jiangsu Provincial People's Hospital, Jiangsu Province, Nanjing 210029, China; Min Yan, MD, Principal Investigator — Henan Cancer Hospital; Yanxia Shi, MD, Principal Investigator — Sun Yat-sen University Cancer Hospital
Locations (5):
- China (5):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Hospital, Guangzhou, Guangdong
  - Second Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided